CLINICAL TRIAL: NCT06022562
Title: Effects of Gender-affirming Hormone Therapy on the Psychosocial and Quality of Life of Transgender People: A Prospective Cohort Study
Brief Title: Effects of Gender-affirming Hormone Therapy on Transgender People
Status: Completed | Type: Observational
Sponsor: National Taiwan University (Other)
Responsible Party: Principal Investigator, Piao-Yi Chiou, Associate Professor, National Taiwan University
Other Study IDs: 202302HM008
Record Dates: First submitted 2023-08-25; First posted 2023-09-05 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Gender Dysphoria
Keywords: depression; gender-affirming hormone therapy
MeSH Terms: conditions — Gender Dysphoria; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- With gender-affirming hormone therapy: With gender-affirming hormone therapy
- Without gender-affirming hormone therapy: Without gender-affirming hormone therapy

SUMMARY:
This prospective cohort study aims to assess the impact of gender-affirming hormone therapy (GAHT) on transgender individuals' physical, psychological, social, and quality of life aspects. Based on gender minority stress theory, the research recruits 150 individuals each of those starting GAHT and those not yet undergoing it. Data collection involves questionnaires and physiological measurements. Statistical analyses will explore correlations and group differences. Findings can guide transgender individuals considering hormone therapy and enhance care guidelines to improve their overall well-being.

DETAILED DESCRIPTION:
The willingness and proportion of transgender persons diagnosed with gender dysphoria to receive gender-affirming hormone therapy (GAHT) is relatively high, so as to conform to their internal gender identity. However, there are limited studies on the prospectively observation of the influences and effectiveness of GAHT on physical, psychological, social and quality of life of transgender people. This study is a cross-sectional research prospective cohort study design, and the research framework is developed based on gender minority stress theory. It is expected to recruit a group of 150 transgender people, including trans male, trans female, and non-binary person, who have just started using GAHT, and a group of 150 who has not yet received GAHT. The data collection time is about 40-50 minutes each time. The questionnaires will be applied to collect basic demographic information, basic hormonal information, body changes, body image, sexual wellbeing, sexual risk, depression, social support, and quality of life. The instruments will be applied to measure participants' physiological parameters, including weight, body fat, and muscle mass, hand grip strength, and blood pressure. In the statistical part, correlation and regression will be used to analyze the degree of correlation between variables, and multivariate analysis of covariance will be used to detect whether there was a significant difference between the variables of the two groups. A well understanding of the experiences and reactions of transgender people receiving hormone therapy can provide a reference for transgender people before deciding to accept hormone therapy, and can be used as an important reference for formulating care guidelines for gender-affirming hormone therapy to improve the care quality for the gender minority population.

ELIGIBILITY:
Inclusion Criteria:

* transgender

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: transgender
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Transgender Congruence Scale | 1 year
  Participants rated this 15 items scale on a 5-point Likert-type scale (i.e., 1 = strongly disagree, 2 = somewhat disagree, 3 = neither agree nor disagree, 4 = somewhat agree, 5 = strongly agree). Four of the 15 items were designed to be reverse-scored. Item responses were averaged, with higher scores indicating a higher level of congruence. So the maximum and minimum values of this scale are 75 and 15.
Gender Affirming Hormone Treatment Physical Symptoms Assessment Scale | 1 year
  Participants rated this 17 items scale on a 4-point Likert-type scale. With higher scores indicates a higher level.
Sexual Risk Survey (SRS) Items | 1 year
  Participants rated this 23 items. This questionnaire inquires about the frequency of subjects' experiences with each sexual risk. A higher frequency indicates a greater level of risk.
Short Sexual Well Being Scale | 1 year
  Participants rated this 5 items scale on a 7-point Likert-type scale. With higher scores indicates a higher level.
Transgender individual Quality of Life | 1 year
  Participants rated this 23 items scale on a 4-point Likert-type scale. With higher scores indicates a higher level.
Beck Depression Inventory-II | 1 year
  The BDI-II, or Beck Depression Inventory-II, is a widely used self-report assessment tool for measuring the severity of depression. It consists of 21 multiple-choice questions or items. Of these 21 items, 13 are scored in the direction of increasing depression severity, while the remaining 8 are reverse-scored to assess positive attributes.
  The possible score range on the BDI-II is from 0 to 63, with higher scores indicating more severe depressive symptoms.
Multidimensional Perceived Social Support Scale | 1 year
  The Multidimensional Perceived Social Support Scale (MPSSS) is a self-report questionnaire designed to assess an individual's perception of the level of social support they receive. It measures support from various sources, such as family, friends, and significant others, and evaluates different dimensions of support, including emotional, instrumental, and informational support. Participants rated this 13 items scale on a 4-point Likert-type scale with 4 different social related group. With higher scores indicates a higher level.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, College of Medicine, School of Nursing, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided